CLINICAL TRIAL: NCT04587622
Title: A Phase 1, Open-label, Single-dose, Parallel-group Study to Evaluate the Systemic Pharmacokinetics of Icenticaftor in Participants With Mild, Moderate, or Severe Hepatic Impairment Compared to Matched Healthy Control Participants
Brief Title: Pharmacokinetic Study of Icenticaftor in Participants With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQBW251A2104
Record Dates: First submitted 2020-09-29; First posted 2020-10-14 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Hepatic Failure
Keywords: Hepatic impairment; Child-Pugh classification; Icenticaftor; QBW251
MeSH Terms: conditions — Liver Failure | interventions — icenticaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 - Healthy subjects with normal hepatic function (Experimental): Healthy subjects with normal hepatic function - Control
  Interventions: Drug: Icenticaftor
- Group 2 - Mild Hepatic Impairment (Experimental): Mild hepatic impairment: Child-Pugh A (Score 5-6)
  Interventions: Drug: Icenticaftor
- Group 3 - Moderate Hepatic Impairment (Experimental): Moderate hepatic impairment: Child-Pugh B (Score 7-9)
  Interventions: Drug: Icenticaftor
- Group 4 - Severe Hepatic Impairment (Experimental): Severe hepatic impairment: Child-Pugh C (Score 10-15)
  Interventions: Drug: Icenticaftor

INTERVENTIONS:
Drug: Icenticaftor — Single oral dose of 300 mg of icenticaftor (QBW251)
  Other Names: QBW251

SUMMARY:
The primary purpose of this study is to evaluate the effect of hepatic impairment on the systemic pharmacokinetics, safety, and tolerability of icenticaftor in participants with varying degrees of hepatic impairment.

DETAILED DESCRIPTION:
This is a Phase 1, multi-center study with parallel groups. The study employs a single-dose, open-label design in subjects with mild, moderate, or severe hepatic impairment along with matched healthy control subjects with normal hepatic function. Subjects with normal hepatic function will be matched with subjects with hepatic impairment for gender, age (± 10 years), body weight (± 15%), and smoking status (smoker or non-smoker).

Up to a total of 48 participants will be enrolled in this study (approximately 8 in each mild [Child-Pugh A], moderate [Child-Pugh B], severe hepatic impairment [Child-Pugh C] groups), and up to 24 healthy control subjects). Each participant will receive a single oral dose of 300 mg of icenticaftor (QBW251) on Day 1 under fasting conditions.

The study is comprised of an up to 28-day screening period (Days -28 to -1), a baseline evaluation (Day -1) prior to treatment on Day 1, and a follow-up period of 7 days for pharmacokinetics (PK) sample collection (pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose). A safety follow-up contact will be done 30 days after administration of the study drug.

The primary purpose of this study is to evaluate the effect of hepatic impairment on the systemic PK, safety, and tolerability of icenticaftor in participants with varying degrees of hepatic impairment.

ELIGIBILITY:
All Participants:

Inclusion Criteria:

* Male and non-child bearing potential female participants, 18 to 75 years of age (inclusive) at Screening.
* Participants must weigh at least 50.0 kg and must have a body mass index (BMI) within the range of 18.0 to 38.0 kg/m2, inclusive, at Screening.
* Must be a non-smoker or agree to smoke no more than 5 cigarettes (or equivalent) per day from Screening until the End of Study. Participants must maintain the same smoking status throughout the study (i.e. smoker or non smoker).

Exclusion Criteria:

* Use of other investigational drugs within 5 half-lives prior to dosing of study treatment, or within 30 days, whichever is longer; or longer if required by local regulations.
* Are taking medications prohibited to be taken with the study treatment
* Known history of, or current clinically significant arrhythmias. Have clinically significant ECG abnormality or history of long-QT syndrome or whose QT interval corrected by Fridericia's formula (QTcF) is prolonged (> 480 msec) at Screening. Participants having myocardial infarction ≥ 5 years ago are eligible to participate.
* Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection.

Healthy Participants:

* Each participant must match in age (± 10 years), gender, weight (± 15%), and smoking status to participants in Group 2, 3, or 4.
* Seated vital signs must be within the following ranges at Screening and Baseline:
* Body temperature, 35.0 to 37.5°C, inclusive.
* Systolic blood pressure, 89 to 149 mmHg, inclusive.
* Diastolic blood pressure, 50 to 89 mmHg, inclusive.
* Pulse rate, 40 to 90 bpm, inclusive.
* Participants must be in good health as determined by medical history, physical examination, ECG, and clinical laboratory tests at Screening.

Exclusion Criteria:

* Liver disease or liver injury as indicated by abnormal liver function tests.
* Chronic infection with HBV or HCV.
* History or presence of impaired renal function.

Hepatic Impairment Participants:

Inclusion Criteria:

* Seated vital signs must be within the following ranges at Screening and Baseline:
* Body temperature, 35.0 to 37.5°C, inclusive.
* Systolic blood pressure, 89 to 159 mmHg, inclusive.
* Diastolic blood pressure, 50 to 99 mmHg, inclusive.
* Pulse rate, 50 to 99 bpm, inclusive.
* Hepatic impairment as defined by the Child-Pugh classification for severity of liver disease

Exclusion Criteria:

* Have severe complications of liver disease within the preceding 3 months of Screening.
* Emergency room visit or hospitalization due to liver disease within the preceding 3 months of Screening.
* Have received liver transplant at any time in the past.
* Have encephalopathy Grade 3 or worse within 28 days prior to dosing of study treatment.
* Have acute hepatitis B (HBV) or hepatitis C (HCV) infection.
* Clinically significant abnormal findings in physical examination or clinical laboratory evaluations not consistent with known liver disease.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Maximum observed icenticaftor plasma concentration (Cmax) after single oral dose | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Icenticaftor plasma concentrations will be determined by a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) method. Cmax of icenticaftor will be determined with Phoenix WinNonlin (Version 6.4 or higher).
Area under the plasma concentration-time curve from time zero to the last measurable concentration sampling time (AUClast) of icenticaftor after single oral dose | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  AUClast of icenticaftor will be determined using non-compartment methods with Phoenix WinNonlin (Version 6.4 or higher). The linear trapezoidal rule will be used for AUClast calculation.
Area under the plasma concentration-time curve from time zero to infinity (AUCinf) of icenticaftor after single oral dose | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  AUCinf of icenticaftor will be determined using non-compartment methods with Phoenix WinNonlin (Version 6.4 or higher). The linear trapezoidal rule will be used for AUCinf calculation.
Time to reach maximum icenticaftor plasma concentration (Tmax) after single oral dose | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Icenticaftor plasma concentrations will be determined by a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) method. Tmax of icenticaftor will be determined with Phoenix WinNonlin (Version 6.4 or higher).
Apparent plasma clearance (CL/F) of icenticaftor after single oral dose | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  CL/F of icenticaftor will be determined using non-compartment methods with Phoenix WinNonlin (Version 6.4 or higher).
Apparent volume of distribution during terminal phase (Vz/F) of icenticaftor after single oral dose | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Vz/F of icenticaftor will be determined using non-compartment methods with Phoenix WinNonlin (Version 6.4 or higher).
Elimination half-life (T1/2) of icenticaftor after single oral dose | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  T1/2 of icenticaftor will be determined using non-compartment methods with Phoenix WinNonlin (Version 6.4 or higher). Regression analysis of the terminal plasma elimination phase will be used for T1/2 calculation.

SECONDARY OUTCOMES:
Plasma protein binding free fraction (unbound fraction [fu]) of icenticaftor | 3 hours post-dose
  The free fraction in plasma fu of icenticaftor will be evaluated at 3 hours post-dose using equilibrium dialysis method.
Cmax of unbound icenticaftor (Cmax,u) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Icenticaftor Cmax,u will be calculated as Cmax*fu.
AUClast of unbound icenticaftor (AUClast,u) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Icenticaftor AUClast,u will be calculated as AUClast*fu.
AUCinf of unbound icenticaftor (AUCinf,u) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Icenticaftor AUCinf,u will be calculated as AUCinf*fu.
CL/F of unbound icenticaftor (CL/F,u) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
  Icenticaftor CL/F,u will be calculated as CL/F/fu.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CQBW251A2104 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18083
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1570